CLINICAL TRIAL: NCT00077064
Title: A Phase II Randomized Trial With Captopril In Patients Who Have Received Radiation Therapy +/- Chemotherapy For Stage II-IIIB Non-Small Cell Lung Cancer, Stage I Central Non-Small Cell Lung Cancer, Or Limited-Stage Small-Cell Lung Cancer
Brief Title: Captopril in Treating Patients With Non-Small Cell Lung Cancer or Limited-Stage Small Cell Lung Cancer That Has Been Previously Treated With Radiation Therapy With or Without Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to unmet accrual/randomization goals
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG-0123; CDR0000315569; RTOG-L-0123
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Results first posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Lung Cancer; Pulmonary Complications; Radiation Fibrosis
Keywords: radiation fibrosis; pulmonary complications; limited stage small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Radiation Fibrosis Syndrome; Carcinoma, Non-Small-Cell Lung | interventions — Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Clinical observation
- Captopril (Experimental): Captopril
  Interventions: Drug: captopril

INTERVENTIONS:
Drug: captopril — Captopril 12.5 mg t.i.d. for first two weeks, increased to 25 mg t.i.d. for the second two weeks of therapy. Thereafter, the dose will be increased to 50 mg t.i.d. for the remainder of the one-year of therapy (52 total weeks of drug administration).
  Arms: Captopril

SUMMARY:
RATIONALE: Captopril is a drug that may be able to decrease side effects caused by radiation therapy, and may improve the quality of life of patients with non-small cell lung cancer or limited-stage small cell lung cancer.

PURPOSE: This randomized phase II trial is studying how well captopril works in decreasing side effects and improving the quality of life in patients who have received radiation therapy with or without chemotherapy for stage I, stage II, or stage IIIB non-small cell lung cancer or limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of captopril on the incidence of pulmonary damage at 12 months after radiotherapy with or without chemotherapy in patients with stage II-IIIB non-small cell lung cancer, stage I central non-small cell lung cancer, or limited stage small cell lung cancer.
* Compare the quality of life of patients treated with captopril vs patients who undergo post-radiotherapy observation only.
* Determine the persistence of captopril's effect on pulmonary toxicity in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, total lung irradiated (< 25% vs 25-37% vs more than 37%), prior surgery (yes vs no), and prior chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral captopril 3 times daily for 1 year in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo observation only for 1 year. Quality of life is assessed at baseline and at months 3, 6, 12, and 18.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 205 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following histologically or cytologically confirmed diagnoses:

  * Stage II-IIIB non-small cell lung cancer (NSCLC)
  * Stage I central NSCLC

    * No peripheral coin lesions
  * Limited stage small cell lung cancer

    * Nonmetastatic disease that is receiving radiotherapy and the target is confined to a single radiotherapy treatment area
* Planning to receive radiotherapy

  * At least 45 Gy to be delivered to the target volume
  * More than 25% of total lung volume to receive > 20 Gy if receiving radiotherapy alone

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Hematopoietic

* Absolute granulocyte count greater than 1,000/mm^3
* Platelet count greater than 75,000/mm^3
* Hemoglobin greater than 9.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin less than 1.5 mg/dL
* Serum glutamate oxaloacetate transaminase (SGOT) less than 2 times normal

Renal

* Blood urea nitrogen (BUN) less than 25 mg/dL
* Creatinine less than 1.6 mg/dL
* Urine protein less than 10 mg/dL
* Urine glucose negative

Cardiovascular

* Systolic blood pressure greater than 110 mm Hg
* Diastolic blood pressure greater than 60 mm Hg

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Sodium normal
* Potassium normal
* No collagen vascular disease (e.g., lupus or scleroderma)

  * Rheumatoid arthritis allowed
* No known hypersensitivity to ACE inhibitors

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Induction or concurrent chemotherapy allowed either during radiotherapy or during therapy with captopril
* No concurrent methotrexate

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Prior pulmonary lobectomy or segmentectomy allowed

  * No prior pneumonectomy

Other

* No concurrent angiotensin-converting enzyme (ACE) inhibitors or angiotensin II receptor antagonists for hypertension or congestive heart failure
* No concurrent lithium
* No concurrent procainamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2003-06; Primary Completion 2008-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Small, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (87):
- United States (87):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - General Robert Huyser Cancer Center at David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Cancer Treatment Center for Southern Kentucky, Bowling Green, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - Trinity CancerCare Center, Minot, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - CCOP - Greenville, Greenville, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were registered within 7 days prior to start of radiation therapy(RT) or during RT up to 48 hours prior completion of RT. They were randomized to captopril or observation within 48 hours prior to completion of RT. Eighty-one patients were registered, 48 did not continue to treatment assignment, 33 were randomized.
Groups:
- Clinical Observation: Clinical observation
- Captopril: Captopril: 50 mg t.i.d.
Period: Overall Study
Arm/Group | Clinical Observation | Captopril
Started | 17 | 16
Completed | 17 (Randomized eligible subjects are considered to have completed the study.) | 10 (Randomized eligible subjects are considered to have completed the study.)
Not Completed | 0 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Patient refusal | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Captopril | Total
Number analyzed (Participants) | 17 | 10 | 27
Age, Continuous [Median (Full Range); unit: years] | 67 [42 to 87] | 64 [46 to 75] | 65 [42 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Therapy-induced Lung Toxicity
Description: Incidence of Grade 2+ radiation-induced pulmonary toxicity within 1 year after completion of radiation. Assuming that the incidence of pulmonary toxicity would be 50%, based on Fisher's exact test with a one-sided significance level of 0.05,168 randomized patients would be required to have 80% statistical power to detect a 40% relative reduction (from 50% to 30%) in the incidence of pulmonary toxicity while receiving captopril. Assuming that 15% of cases would not continue to the randomization stage and 5% of patients would be found ineligible, the target sample size was 205 patients. Given the actual sample size, power would be 25% and therefore p-values were not reported.
Time Frame: Once all patients have been followed for at least 12 months
Population: Randomized eligible patients who started study drug treatment and were followed for one year after completion of radiation treatment or experienced radiation-induced pulmonary toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation | Captopril
Number analyzed (Participants) | 13 | 7
percentage of participants | 23 [11 to 35] | 14 [4 to 24]

2. Secondary Outcome: Correlation of Lung Toxicities With Biochemical Markers
Description: Biomarker data will not be generated from these tissue specimens, therefore this analysis will not take place.
Time Frame: Once all patients have been followed for at least 12 months
Arm/Group | Clinical Observation | Captopril
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Correlation of Quality of Life With Late Effects as Measured by European Organization for Research and Treatment of Cancer (EORTC) C-30 or EORTC Lung Cancer Module (LC-13)
Description: Only 2 patients have the required data- only 1.2% of the planned enrollment and 2.5% of the actual enrollment- which is extremely problematic as this data cannot be generalized, leads to selection bias, and is not representative of the patient population. Therefore the analysis was not conducted.
Time Frame: Baseline to 18 months post treatment
Population: Eligible patients with late effect and baseline and 12-month EORTC data
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Observation | Captopril
Number analyzed (Participants) | 2 | 0
Participants | NA — Insufficient number of participants with data collected to derive a correlation |

4. Secondary Outcome: Persistence of Pulmonary Toxicity at 2 Years After Completion of Study Treatment
Description: Patients who experienced a Grade 2+ radiation-induced pulmonary toxicity within 1 year after completion of radiation were assessed to determine if the toxicity persisted for 2 years.
Time Frame: 2 years from completion of study treatment
Population: Randomized patients who received study drug treatment and experienced lung toxicity at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Observation | Captopril
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Description: Adverse events reported for all eligible randomized patients who were randomized to captopril or observation. Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE).
Arm/Group | Clinical Observation | Captopril
Serious Adverse Events (participants affected / at risk) | 8/17 | 8/10
Other Adverse Events (participants affected / at risk) | 8/17 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clinical Observation (N=17) | Captopril (N=10)
Cardiac General - Other: (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Esophageal pain (Gastrointestinal disorders) | 1 | 1
Esophageal stenosis acquired (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oseophagitis NOS (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Disease progression NOS (General disorders) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Urinary tract NOS (Infections and infestations) | 0 | 1
Vessel injury-vein: SVC (Injury, poisoning and procedural complications) | 1 | 0
Lymphopenia (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary/upper respiratory - Other: (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension NOS (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clinical Observation (N=17) | Captopril (N=10)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Oseophagitis NOS (Gastrointestinal disorders) | 1 | 1
Salivary gland disorder NOS (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 5 | 6
Infection - Other: (Infections and infestations) | 1 | 0
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Metabolic/laboratory - Other: (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3
Headache (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1

LIMITATIONS AND CAVEATS:
The study stopped accrual early due to unmet accrual/randomization goals: 81 accrued of 205 planned, 33 randomized of 168 planned. Statistical testing of primary outcome measure not done due to low power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.